CLINICAL TRIAL: NCT02439866
Title: The Effect of High Dose Steroid and Normobaric Oxygen Therapy on Recent Onset Non-arteritic Anterior Ischemic Optic Neuropathy(NAION); a Randomized Clinical Trial
Brief Title: Outcomes of Steroid and Oxygen Therapy Versus Placebo Therapy in Non-arteritic Anterior Ischemic Optic Neuropathy
Acronym: NAION
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Shahid Beheshti Medical University, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 93222
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2014-01

CONDITIONS: NAION( Non-arteritic Anterior Ischemic Optic Neuropathy)
MeSH Terms: interventions — Masks

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- prescription placebo (Placebo Comparator): control Group consisted of 30 patients who received gelatinous capsules filled with sugar as placebo
  Interventions: Drug: placebo
- prescription Intravenous methylprednisolone (Active Comparator): Group 2 or steroid consisted of 30 patients received methylprednisolone (Solu-Medrol, Pharmacia Pharmaceutical Company, Belgium) 500 mg twice a day for 3 days followed by 2 weeks of oral prednisolone 1mg/kg/day
  Interventions: Drug: Intravenous methylprednisolone
- prescription normobaric oxygen with face mask (Active Comparator): Thirty patients in group 3 or oxygen received 100% normobaric oxygen with face mask in sitting position, at a flow rate of 5 liters per minute for 1 hour twice a day for two weeks
  Interventions: Drug: normobaric oxygen with face mask

INTERVENTIONS:
Drug: placebo — gelatinous capsules filled with sugar as placebo
  Arms: prescription placebo
Drug: Intravenous methylprednisolone — Intravenous methylprednisolone (Solu-Medrol, Pharmacia Pharmaceutical Company, Belgium) 500 mg twice a day for 3 days followed by 2 weeks of oral prednisolone 1mg/kg/day (Prednisolone Fort; Sina Daroo, Iran
  Arms: prescription Intravenous methylprednisolone
Drug: normobaric oxygen with face mask — normobaric oxygen100% with face mask in sitting position, at a flow rate of 5 liters per minute for 1 hour twice a day for two weeks
  Arms: prescription normobaric oxygen with face mask

SUMMARY:
Patients diagnosed with NAION within 14 days of onset were included. Patients were randomized into 3 groups. Group 1 or control consisted of 30 patients who received gelatinous capsules filled with sugar as placebo. Group 2 or steroid consisted of 30 patients received methylprednisolone (Solu-Medrol, Pharmacia Pharmaceutical Company, Belgium) 500 mg twice a day for 3 days followed by 2 weeks of oral prednisolone 1mg/kg/day. Thirty patients in group 3 or oxygen received 100% normobaric oxygen with face mask in sitting position, at a flow rate of 5 liters per minute for 1 hour twice a day for two weeks Functional and structural outcomes were assessed at 1 and 6 months following treatment. Best corrected visual acuity was the main outcome measure, and mean deviation index of visual field test and peripapillary retinal nerve fiber layer thickness were secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recent onset ( within 2 weeks) of non-arteritic ischemic optic neuropathy

Exclusion Criteria:

* the presence of glaucoma, or any other ocular, neurologic, or systemic disease that may influence visual acuity and visual field; abnormal results in laboratory assessments, including an abnormally elevated erythrocyte sedimentation rate and positive serum C-reactive protein;
* a history of previous ocular surgery;
* a history of prior treatment of any type for NAION;
* systemic condition such as diabetes mellitus and poorly controlled hypertension

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity using Snellen chart | until 6 months
  Snellen chart

SECONDARY OUTCOMES:
Visual field mean deviation index using the Humphrey Visual Field Analyzer | until 6 months
  the Humphrey Visual Field Analyzer (HFA; model 750; Carl Zeiss Meditec, Inc., Dublin, California, USA)

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran, Iran